CLINICAL TRIAL: NCT01555840
Title: "EVALUATION CLINIQUE D'UNE CAPSULE A GUIDAGE MAGNETIQUE POUR L'EXPLORATION GASTRIQUE "Capsule Dirigée Versus Gastroscopie à Haute Définition""
Brief Title: Comparative Study of the Magnetically Guided Capsule Endoscopy Versus High Definition Gastroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Institute Arnault Tzanck, France (Other); Centre Hospitalier Universitaire de Nice (Other); Keio University (Other); Showa University Northern Yokohama Hospital, Japan (Unknown); The Jikei University School of Medicine, Japan (Unknown); Olympus Corporation (Industry); Siemens AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2010-A01442-37(AFSSAPS)
Record Dates: First submitted 2012-03-07; First posted 2012-03-15 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Gastric Focal Lesion
Keywords: Magnetically guided capsule endoscopy (MGCE); Gastroscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients requiring upper GI endoscopy (Other): patients with upper abdominal complaints requiring upper GI endoscopy
  Interventions: Device: Magnetically Guided Capsule (MGCE)

INTERVENTIONS:
Device: Magnetically Guided Capsule (MGCE) — "a) MGCE capsule The MGCE capsule is custom-made for observation of the stomach. It is 31 mm in length and 11 mm in diameter and equipped with two image sensors.
  It contains a permanent magnet to enable magnetic guidance in the stomach by magnetic field." "b) Guidance system The magnet guidance system is custom-made to guide the MGCE capsule inside the stomach. It has a footprint of 1m× 2m and generates a very low level magnetic fields." c) Conventional gastroscope

SUMMARY:
A capsule steered by magnetic field force developed by Siemens and Olympus has recently been evaluated in a pilot series in man with encouraging results (Rey JF, Ogata H, Hosoe N, Ohtsuka K, Ogata N, Ikeda K, Aihara H, Pangtay I, Hibi T, Kudo S, Tajiri H. Feasibility of stomach exploration with a guided capsule endoscope. Endoscopy. 2010;42:541-5. Epub 2010 Jun 30.18). This blinded prospective study investigates the accuracy of the magnetically guided capsule (MGCE) compared to gastroscopy in patients with focal lesions and / or gastric symptoms and indication for upper GI Endoscopy.

DETAILED DESCRIPTION:
The sudy takes place in a private hospital (Institute Arnault Tzanck, St. Laurent du Var) with an annual number of 4000 upper GI endoscopies. Patients will be recruited from this center and from the cooperating Department of Gastroenterology at the University of Nice by about half. After given written informed consent at least 24 hours prior the examination patients are included into the study. The examiners are blinded to the patients origin.

Participants will be recruited in two groups A) enriched population group (n=50): In both institutions, patients presenting for upper GI endoscopy with suspected or diagnosed focal lesions as follows; gastric tumors, submucosal tumor, gastric ulcer, polyp a)adenoma, b)hyperplastic polyp or angioectasia,ulcers for diagnostic confirmation, follow-up or planning of therapy will be informed and asked to participate in the study.

B) standard gastroscopy group (n=150): consecutive patients without prior gastroscopy presenting with the main indications reflux, upper abdominal complaints, anemia and anorexia. Here, recruitment is based on presenting symptoms.

6 endoscopists experienced in upper GI endoscopy (> 1000 examinations) and specifically trained in capsule gastroscopy (simulator, 10 gastric capsule cases) will perform capsule gastroscopy. 2 well trained endoscopists (> 1000 upper GI endoscopies), different from the capsule gastroscopists will perform subsequent gastroscopies. They receive standard information about gastroscopy indication from a list of indications. They are accompanied by a study nurse who knows patient details but ascertains examiner blindness and takes care of secondary unblinding during gastroscopy.

Gastroscopy is always performed after MGCE in this study with a maximum delay of 1 day but a minimum delay of 4 h due to water filling of the stomach with the capsule examination.

The study is a comparative study of capsule gastroscopy accuracy with conventio¬nal gastroscopy serving as gold standard as described above. Disease prevalence is enriched to include 25-30% of significant pathology such as tumors and ulcers. Confidence intervals will be calculated, e.g. for a disease prevalence of about 30% and 200 study cases, a sensitivity of 85% will have a 95% CI of 73-93%. Cross tabulation of the results of the index tests (including indeterminate and missing results) will be performed by the results of the reference standard. Study statistics will be done by Prof. Dr. Karl Wegscheider, University Hospital Hamburg/Eppendorf.

All patient data will be collected at Institut Arnault Tzanck in St. Laurent du Var. Data will be analyzed in pseudonymity way (code, age, sex) at the University of Hamburg. Original data will be stored for 10 years at Institut Arnault Tzanck in St. Laurent du Var

ELIGIBILITY:
Inclusion Criteria:

* Patients with gastric focal lesions (Group A)
* Patients with gastric symptoms and indicated for Upper GI endoscopy (Group B)
* Age of 18 years to 75 years"

Exclusion Criteria:

* Patients with dysphagia or symptoms of gastric outlet obstruction
* Patients with suspected or known intestinal stenoses
* Overt GI bleeding
* Known large and obstructing tumors of the upper GI tract
* Patients after upper GI surgery or abdominal surgery altering GI anatomy
* Patients under full anticoagulation
* Patient in poor general condition (ASA III/IV)
* Patients with claustrophobia
* Patients using equipment that may be affected by radio transmission
* Patients using equipment that may be affected by magnetic field
* Pregnancy or suspected pregnancy "

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Accuracy of magnetically guided capsule endoscopy (MGCE) as compared to unblinded gastroscopy in the diagnosis of focal lesions. | 2 days
  To evaluate the accuracy of MGCE, which is performed by the first examiner. After the MGCE examination, conventional gastroscopy is performed by the second examiner and then the results of the two studies are compared.

SECONDARY OUTCOMES:
Accuracy of capsule endoscopy in the diagnosis of diffuse and minor lesions | 2 days
  - Accuracy of capsule endoscopy in the diagnosis of diffuse and minor lesions [ Time Frame: within 2 days ] [ Designated as safety issue: No ]
Examination times of capsule and conventional gastroscopy | 1 hour
  Examination times of capsule and conventional gastroscopy
Patient acceptance of capsule gastroscopy and conventional gastroscopy | 2 days
  Patient acceptance of capsule gastroscopy and conventional gastroscopy
  * After the two examinations are finished, patients fill out the questionnaire.
Adverse events of both procedures | 14 days
  Adverse events of both procedures

CONTACTS AND LOCATIONS:
Overall Officials: J F Rey, MD, Principal Investigator — Institut Arnault Tzanck, St. Laurent du Var, France
Locations (1):
- Institut Arnault Tzanck , Avenue du Docteur Maurice Donat, Saint-Laurent-du-Var, Cote Azur, France

REFERENCES:
- [Background] Rey JF, Ogata H, Hosoe N, Ohtsuka K, Ogata N, Ikeda K, Aihara H, Pangtay I, Hibi T, Kudo SE, Tajiri H. Blinded nonrandomized comparative study of gastric examination with a magnetically guided capsule endoscope and standard videoendoscope. Gastrointest Endosc. 2012 Feb;75(2):373-81. doi: 10.1016/j.gie.2011.09.030. Epub 2011 Dec 9. PMID 22154417
- [Background] Rey JF, Ogata H, Hosoe N, Ohtsuka K, Ogata N, Ikeda K, Aihara H, Pangtay I, Hibi T, Kudo S, Tajiri H. Feasibility of stomach exploration with a guided capsule endoscope. Endoscopy. 2010 Jul;42(7):541-5. doi: 10.1055/s-0030-1255521. Epub 2010 Jun 30. PMID 20593331
- [Result] Denzer UW, Rosch T, Hoytat B, Abdel-Hamid M, Hebuterne X, Vanbiervielt G, Filippi J, Ogata H, Hosoe N, Ohtsuka K, Ogata N, Ikeda K, Aihara H, Kudo SE, Tajiri H, Treszl A, Wegscheider K, Greff M, Rey JF. Magnetically guided capsule versus conventional gastroscopy for upper abdominal complaints: a prospective blinded study. J Clin Gastroenterol. 2015 Feb;49(2):101-7. doi: 10.1097/MCG.0000000000000110. PMID 24618504